CLINICAL TRIAL: NCT05595304
Title: Evaluation of the Impact on General Functionality of the Application of a Protocol of Immediate Prosthetic Functionalization in Patients With Deficient Removable Prostheses, Compared With the Conventional Treatment That is Delivery at the Secondary Level of the Health System to People Over 70 Years
Brief Title: Impact on General Functionality of an Immediate Prosthetic Functionalization Protocol in People Over 70 Years of Age With Deficient Removable Prostheses
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gerardo F Fasce Pineda, MD (Other Government)
Responsible Party: Sponsor-Investigator, Gerardo F Fasce Pineda, MD, Head of Geriatrics - Hospital Clinico Universidad de Chile, Comisión Nacional de Investigación Científica y Tecnológica
Organization: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SA20I0052
Record Dates: First submitted 2022-10-20; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Removable Dental Prosthesis; Dental Restoration; Elderly; Functional Status

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Functionalization (Experimental): Prosthesis repairment: prosthetic reline and occlusal stabilization through repair of missing pieces and recovery of occlusal contacts and follow up with conventional prosthesis treatment
  Interventions: Procedure: prosthetic refunctioning
- control (Active Comparator): conventional prosthetic treatment (new prosthesis)
  Interventions: Procedure: conventional prosthetic treatment

INTERVENTIONS:
Procedure: prosthetic refunctioning — Active treatment followed by regular interventions
  Arms: Oral Functionalization
Procedure: conventional prosthetic treatment — new prosthesis
  Arms: control

SUMMARY:
Title: Evaluation of the impact on general functionality of the application of an immediate prosthetic functionalization protocol, in patients with deficient removable prostheses, compared with the conventional treatment that is delivered at the secondary level of the health system, to people over 70 years of age.

Introduction: Sarcopenia and malnutrition are closely involved in frailty. To prevent them it is important to assess oral function. "Oral fragility" manifests with specific signs or symptoms, among which are loss of occlusion due to tooth loss and chewing difficulty. To recover from it, it is important to restore function by placing a dental prosthesis in the event of tooth loss. In Chile, a large percentage of patients who are referred to secondary care to perform new prosthetic treatment, lives in conditions of less oral functionality and enters waiting lists that can take years, with a silent impact on general functionality. Falls are a public health problem with a significant economic cost, being the second cause of death worldwide. One of the causes is sarcopenia and it has been studied that the decrease in the number of teeth and the occlusal posterior support region may be risk factors for decreased gait speed, an objective measurement of fall risk. It has been studied that the decrease in the number of teeth causes a reduction in: total muscle mass, walking speed and lower quality of life.

Hypothesis: The recovery of immediate functionality in deficient prostheses in patients 70 years of age and older will have a positive and rapid impact on general functionality and on their assessment of oral health related quality of life.

General objective: To evaluate the impact on general functionality of the application of an immediate prosthetic functionalization protocol in patients with deficient removable prostheses, compared with conventional treatment, at the secondary level of the health system, in patients over 70 years of age.

Methodology: randomized, double-blind clinical trial with two groups of 62 patients each: experimental and control. The intervention will consist of recovering prosthetic function in one session, before conventional rehabilitation vs. the control group that will receive conventional rehabilitation. Measurements will include manual grip strength measurements, made with a Jamar dynamometer, timed up and go test, before and after prosthetic treatments and quality of life related to oral health through Ohip 7sp. Descriptive statistics will be applied, through the registration of frequency and contingency tables. To compare hand grip strength, the Pearson's Correlation will be used; for risk of pre and post fall, the t-test will be applied for 2 related samples; for quality of life before and after intervention, Chi2 will be used; changes in grip strength, fall risk and quality of life, between the different groups according to the Eichner index, one-way ANOVA will be applied, for related samples.

Results: A short-term improvement is expected in patients whose functionality will be recovered, which, being a simple technique of competence of the general dentist, could be applied in primary care, without loss of valuable time before attention is achieved, at the secondary level for rehabilitation with new prostheses.

DETAILED DESCRIPTION:
In the public health system, older adults who need new dental prostheses are referred from primary health care to the rehabilitation specialty at the secondary care level. In many cases, they wear old, fractured, non-functional prosthetic devices and enter waiting lists for several months at the hospital level. During that time, they continue a process of oral hypofunction, a stage that gradually progresses to a process of oral dysfunction and decreased systemic function. Once they are called from the secondary level to enter treatment, they must wait for the rehabilitation process time that takes about two months, a period in which they continue with oral hypofunction, a functional pathophysiological condition that closely maintains the negatively impact in nutrition. Our proposal consists of carrying out a dental intervention, competence of the general dentist, when the patient begins the conventional treatment process, once you enter secondary care. This intervention is intended to immediately recover bilateral, homogeneous and simultaneous occlusal contacts, in addition to recovering the prosthetic biomechanical characteristics, by improving prosthetic support, retention and stability. All of this will be made with supplies commonly used in the dental clinic in health services and university teaching clinics. To evaluate the effect that this intervention will have at the muscular level, the patient's manual grip strength and gait speed will be measured, before the intervention and fifteen days later. Subsequently, once the new prostheses have been made, a new measurement will be made. A quality of life survey related to oral health will be applied to both groups, before and after the intervention and treatment. Based on international scientific evidence and on an investigation carried out by this research team (presented at the Chilean National Congress of Geriatrics and Gerontology), between October 2018 and April 2019 in 60 octogenarian older adults not wearing prostheses in whom dental prostheses were built - whose objective was to determine if there was an association between the use of prostheses that return the premolars and molars and the gripping force of the hand. Hand tightening force was measured before and 15 days after prosthetic rehabilitation with a manual hydraulic dynamometer (Jamar MR). For the cohort in study the use of prostheses increased the gripping force of the hand by a statistically significant value. This research aims to be a contribution for the Chilean population and for geriatrics, since the immediate recovery of oral functionality will eliminate a risk factor in older people, reducing conditions that increase frailty, which in cases of entering long-term lists is expected to have a greater impact at the systemic level and higher health costs. In some cases, out-of-pocket spending on dental supplies will also be reduced, because by recovering prosthetic biomechanical conditions, older people will not have to invest resources in creams and/or adhesive powders to "improve" prosthetic adhesion. With this, it would also be possible to contribute to the improvement of the quality of life of these patients as a result of the recovery of functions: masticatory and social. It will also allow a better integration of dentists into the multidisciplinary team in the care model proposed by the Health Ministry and will allow the development and implementation of a care protocol in primary health care, considering that the intervention will contemplate actions that are the responsibility of general dentists.

Without the development of this research, care system will maintain its long waits for this age group for treatment, a situation that will continue to increase considering that global projections related with a greater increase in older inhabitants, and also of the costs already described.

ELIGIBILITY:
Inclusion Criteria:

* 70 or older
* Willingness to participate
* Discharged from Primary Care to the Oral Health Department at Hospital Salvador, Santiago Chile for prosthetic treatment
* With both maxilar an mandibular prosthesis affected
* Eichner groups B3, B4, C1, C2 and C3.

Exclusion Criteria:

* Cognitive impairment (Pfeiffer test classified as moderate or severe)
* Diseases that affect the ability to use facial muscles
* Soft Tissue diseases that affect facial functionality like fibroids

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Handgrip strength | 15-30 days
  measurment in kilograms of handgrip strength. Higher scores mean a better outcome
Falls Risk | 15-30 days
  Measurement of Time up and go test. Measured in seconds. Higher scores mean worse outcomes
Estimation of Quality of Life | 15-30 days
  Use of Oral Health Impact Profile Ultra Short Version (OHIP 7Tsp) survey. Score from 0 to 28, higher scores mean worse outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Salvador, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided